CLINICAL TRIAL: NCT03702166
Title: Network Dysregulation Among Individuals With Comorbid Tinnitus and PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, John Moring, John Moring, PhD, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20180524H; 1KL2TR002646-01 (NIH)
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Results first posted 2020-12-16 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Stress Disorders, Post-Traumatic; Tinnitus
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Tinnitus | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional CPT (Other): This study will examine the effectiveness of Cognitive Processing Therapy (CPT) for the alleviation of PTSD and tinnitus-related distress among individuals with co-morbid PTSD and tinnitus.
  Interventions: Behavioral: Cognitive Processing Therapy (CPT)

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy (CPT) — CPT is a cognitive behavioral treatment for PTSD consisting of 12 one-hour sessions. CPT is delivered in three phases: education, processing, and challenging.
  Other Names: CPT

SUMMARY:
Evaluation of the overlap between tinnitus-related distress and symptoms of Post Traumatic Stress Disorder (PTSD), to identify functional covariance among resting-state networks among individuals with tinnitus and PTSD

DETAILED DESCRIPTION:
The purpose of this study is to characterize tinnitus and PTSD symptomatically, neurobiologically, and causally, applying causal modeling to psychometric and neurofunctional data. We will enroll 30 individuals with both tinnitus and PTSD. Participants will be asked to complete baseline assessments of subjective tinnitus distress, PTSD, depression, and resting-state fMRI at baseline. Individuals with comorbid tinnitus and PTSD who are eligible for the study will receive 12 sessions of Cognitive Processing Therapy (CPT) over a 6- to 15-week period. CPT is a trauma-focused treatment for PTSD that guides individuals on how to recognize and challenge thoughts that are erroneous and dysfunctional. One-month follow-up assessments of tinnitus-related distress, PTSD, depression, and anxiety will be conducted, along with resting-state functional magnetic resonance imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

* Adult military Veterans (age 18-60) who deployed in support of combat operations post-9/11 seeking behavioral health treatment for PTSD and/or tinnitus
* Diagnosis of PTSD determined by the Clinician-Administered PTSD Scale - Interview - Version 5 (CAPS-5)
* Ability to speak and read English
* Meets criteria for tinnitus and considers their tinnitus bothersome, as defined by a score on the Tinnitus Functional Index of 32 or greater

Exclusion Criteria:

* Currently receiving evidence based treatment for PTSD
* Current suicidal ideation severe enough to warrant immediate attention (as determined by the Depressive Symptoms Index- Suicidality Subscale and corroborated by a clinical risk assessment by a credentialed provider
* Psychiatric hospitalization in the last 12 months
* Current and severe alcohol use warranting immediate intervention based on clinical judgment
* Current manic episode or psychotic symptoms requiring immediate stabilization or hospitalization (as determined by the manic and psychosis modules of the MINI)
* Evidence of a moderate or severe traumatic brain injury (as determined by the inability to comprehend the baseline screening questionnaires)
* Neurobiological disorders
* Meniere's disease, temporomandibular joint disorders
* History of seizures
* History of penetrating head trauma or neurosurgery
* Metal objects implanted in the head, ferrous metal filings in the eye
* Inflammation of the brain
* Cardiac pacemaker
* Implanted medical pump or cardiac lines
* Heart disease
* Currently taking certain types of medication for depression or seizures (tricyclic antidepressants or neuroleptics which lower seizure threshold)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Moring, PhD, Principal Investigator — UT Health San Antonio
Locations (1):
- UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Summary results will be shared on ClinicalTrials.gov and will also be shared in publication at study completion.
Supporting Information: Study Protocol, SAP
Time Frame: Study completion

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interventional CPT
Started | 10
Completed (10 participants were started and included in baseline measures, only 8 remained at post-treatment.) | 8
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Interventional CPT
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.3 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Score on Clinician Administered PTSD Scale for the DSM-5 (CAPS-5)
Description: The CAPS-5 is structured interview that assesses the DSM-5 criteria for PTSD. Each item is rated on a severity scale ranging from 0 (Absent) to 4 (Extreme/incapacitating) and combines information about frequency and intensity for each of the 20 symptoms. Total scores range from 0-80 with a lower score indicating less symptoms of PTSD. Subscales were not utilized in analyses.
Time Frame: Baseline and Week 15
Population: Baseline scores pre-treatment included 10 subjects, post-treatment scores included only 8 subjects who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Interventional CPT: This study will examine the effectiveness of Cognitive Processing Therapy (CPT) for the alleviation of PTSD and tinnitus-related distress among individuals with co-morbid PTSD and tinnitus.
  Cognitive Processing Therapy (CPT): CPT is a cognitive behavioral treatment for PTSD consisting of 12 one-hour sessions . CPT is delivered in three phases: education, processing, and challenging.
Arm/Group | Interventional CPT
Number analyzed (Participants) | 10
score on a scale
  Pre-treatment at baseline | 33.10 (7.50)
  Post-treatment at 15 weeks: number analyzed (Participants) | 8
  Post-treatment at 15 weeks | 16.13 (14.49)
Statistical Analysis 1: Comparison: Interventional CPT; Test type: Superiority; p = 0.01, t-test, 1 sided; Multiple t-tests with Bonferroni corrections for multiple comparisons

2. Primary Outcome: Change in Score on the PTSD Check List-5 (PCL-5)
Description: The PCL-5 is a 20-item self-report measure designed to assess PTSD symptoms. The PCL-5 evaluates how much participants have been bothered by PTSD symptoms in the past month (for baseline and follow up assessments) as a result of a specific life event. Each item of the PCL-5 is scored on a five point scale ranging from 0 ("not at all") to 4 ("extremely). Possible total score range is 0-80, with a lower score indicating less PTSD symptoms. Subscales were not utilized in analyses.
Time Frame: Baseline and Week 15
Population: Baseline at pre-treatment included 10 subjects, post-treatment included only 8 subjects who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interventional CPT
Number analyzed (Participants) | 10
score on a scale
  Pre-treatment at baseline | 42.7 (12.25)
  Post-treatment at 15 weeks: number analyzed (Participants) | 8
  Post-treatment at 15 weeks | 17.75 (18.91)

3. Primary Outcome: Change in Score on the Tinnitus Functional Index (TFI)
Description: The TFI has 25 items that are used to calculate eight subscales that address the intrusiveness of tinnitus, the sense of control the patient has, cognitive interference, sleep disturbance, auditory issues, relaxation issues, quality of life, and emotional distress related to tinnitus. The same 25 items are used to calculate the total score, which was used for the purpose of this study. For the total score, the 25 scale items are scored 0-10 (those scored as a percentage are converted to a score of 1-10). Scores are totaled giving a potential range of 0-250 with a higher score indicating that tinnitus interferes more with the subject. The total score is then divided by the number of questions answered to give a mean score. The mean score is multiplied by 10 to provide an overall TFI score within a 0-100 range, where a lower score indicates that the tinnitus does not interfere with the subjects well-being as much.
Time Frame: Baseline and Week 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interventional CPT
Number analyzed (Participants) | 10
score on a scale
  Pre-treatment at baseline | 65.16 (15.97)
  Post-treatment at week 15: number analyzed (Participants) | 8
  Post-treatment at week 15 | 41.95 (24.42)
Statistical Analysis 1: Comparison: Interventional CPT; Test type: Superiority; p = 0.038, t-test, 1 sided; Multiple t-tests, with Bonferroni corrections for multiple comparisons,

4. Primary Outcome: Tinnitus Acceptance Questionnaire (TAQ)
Description: The TAQ captures the extent to which individuals accept their tinnitus, and attempts to avoid or control tinnitus, as well as a patient's ability to pursue valued life activities and meaningful goals regardless of tinnitus. 12 questions are scored from 0 = Never true to 6= Always true. Total scores on the TAQ range from 0-72, with a lower score indicating higher acceptance of symptoms.
Time Frame: Baseline and Week 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interventional CPT
Number analyzed (Participants) | 10
score on a scale
  Pre-treatment at baseline | 35.10 (8.28)
  Post-treatment at 15 weeks: number analyzed (Participants) | 8
  Post-treatment at 15 weeks | 46.88 (13.65)

5. Secondary Outcome: Depression Symptom Index Suicide Subscale (DSI-SS)
Description: The DSI-SS will be used to assess current suicidal ideation. The DSI-SS is a 4-item self-report measure of suicidal ideation that focuses on ideation, plans, perceived control over ideation, and impulses for suicide. Each item is rated on a 4 point scale, and the scores totaled for a potential range of 4-16, where a higher score indicates more severe degrees of suicide ideation.
Time Frame: Baseline and Week 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interventional CPT
Number analyzed (Participants) | 10
score on a scale
  Pre-treatment at baseline | 14.10 (6.59)
  Post-treatment at 15 weeks: number analyzed (Participants) | 8
  Post-treatment at 15 weeks | 7.38 (4.98)
Statistical Analysis 1: Comparison: Interventional CPT; Test type: Superiority; p = 0.031, t-test, 1 sided — Multiple t-tests, with Bonferroni corrections for multiple comparisons

6. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: The PHQ-9 is a widely used and well-validated instrument for measuring the severity of depressive symptoms. It consists of 9 items that assess both affective and somatic symptoms related to depression and depressive disorders that correspond to the diagnostic criteria for Major Depressive Disorder, outlined by the Diagnostic and Statistical Manual of Mental Disorders- 5th Edition (DSM-V, 2013). Each question is rated with a score of 0-3:
  0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day. Scores are the total for the nine questions with a possible range of 0-27, where a lower score indicates minimal depression and a higher score indicates severe depression.
Time Frame: Baseline and Week 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interventional CPT
Number analyzed (Participants) | 10
score on a scale
  Pre-treatment at baseline | 14.10 (6.59)
  Post-treatment at 15 weeks: number analyzed (Participants) | 8
  Post-treatment at 15 weeks | 7.38 (4.98)

ADVERSE EVENTS:
Time Frame: Baseline to 15 weeks
Arm/Group | Interventional CPT
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional CPT (N=10)
Increased irritablilty (Psychiatric disorders) | 2 (2) — Reminder of trauma and impact statement related irritability..
Nightmares (Psychiatric disorders) | 2 (2) — Nightmares related to traumatic event, or unsure of cause.
Adverse memories triggered (Psychiatric disorders) | 1 (1) — Increased memories of the trauma.
Sadness (Psychiatric disorders) | 1 (1) — Increased sadness triggered by thoughts of trauma.
Anxiety (Psychiatric disorders) | 1 (2) — Extreme anxiety during the MRI scan
Sleeplessness (General disorders) | 1 (1) — Lack of sleep due to MRI concerns and back pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT03702166/Prot_SAP_000.pdf